CLINICAL TRIAL: NCT04355897
Title: Convalescent CoVID-19 Plasma in the Treatment of High Risk CoVID-19 Disease
Brief Title: CoVID-19 Plasma in Treatment of COVID-19 Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Dean Kereiakes, Prinicipal Investigator, The Christ Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-23
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Convalescent COVID 19 Plasma (Experimental): Subjects will receive and intravenous infusion of 500 mls of Convalescent COVID 19 Plasma.
  Interventions: Biological: Convalescent COVID 19 Plasma

INTERVENTIONS:
Biological: Convalescent COVID 19 Plasma — Subjects will be transfused intravenously with 500 mls of convalescent COVID 19 plasma

SUMMARY:
The investigatores propose to evaluate intravenous administration of convalescent plasma (CP) obtained from COVID19 survivors in patients requiring hospitalization for symptomatic "high risk" COVID19 disease as reflected by the presence of elevated hsTPN. Supportive data exist for use of convalescent plasma in the treatment of COVID19 and other overwhelming viral illness. Investigators hypothesize that treatment with COVID19 CP will demonstrate salutary effects on COVID19 disease severity/duration, with the primary objective to reduce mortality and a key secondary objective to reduce the requirement for and/or duration of mechanical ventilation. Finally, as the hospital mortality for patients requiring mechanical ventilation is very high (50 to 80%), these patients will be eligible for COVID19 CP treatment as well, even in the absence of elevated hsTPN. Although considerable overlap of these populations has been observed (elevated hsTPN and requirement for mechanical ventilation) there is not 100% redundancy and it is hopeful that COVID19 CP may provide benefit to these critically ill patients.

DETAILED DESCRIPTION:
Coronavirus's are responsible for 15-30% of "common colds" and approximately 2% of the population may be healthy carriers of these viruses. The ongoing SARS CoV-2 pandemic originated in Wuhan, Hubei, China and has spread worldwide. The disease caused by SARS CoV-2 (COVID19) is manifest by fever, fatigue, dry cough, pharyngitis and headache. Although the majority (~80%) COVID19 cases are mild in severity, patients may present with moderate symptoms of dyspnea, tachypnea (~15%) or more severe symptoms (~5-10%) of pneumonia, acute respiratory distress syndrome (ARDS), hypotension, arrythmias and shock(6-9). In addition to the common clinical presentation of respiratory distress, an increasing frequency of cardiovascular manifestations have become evident. These manifestations may be linked to the Angiotensin Converting Enzyme-2 (ACE-2) receptor, a membrane-bound aminopeptidase that has been identified as the functional receptor for SARS CoV-2, which is expressed predominantly in the heart, intestine, kidney and pulmonary alveolar (type 2) cells. Recent data suggest that ~20% of infected subjects may require hospitalization and among patients hospitalized for COVID19, 12-28% will have evidence of myocardial injury (elevated high-sensitivity Troponin: hsTPN) often in association with electrocardiographic (ECG) abnormalities, arrythmias and/or evidence for impaired Left Ventricular contractile function on non-invasive imaging. Indeed, a syndrome of "pseudo-infarction" manifest as ST-segment elevation in the absence of obstructive coronary artery disease has been described. The etiology(s) of myocardial injury may be multifactorial and includes demand ischemia due to critical illness, cytokine storm with atherosclerotic plaque disruption due to overwhelming systemic inflammation and more likely, myocarditis. Indeed, SARS CoV viral RNA along with macrophage infiltration and myocardial cell injury has been detected in autopsied heart samples from patients who succumbed to the SARS outbreak in Toronto. Further, myocardial injury has been directly correlated with both the degree of systemic inflammation (Level of hsCRP) and cardiac dysfunction (level of NT-proBNP). Importantly, myocardial injury was identified to be one of the two most significant, independent predictors (by multi-variable analysis) of hospital death (in addition to ARDS) and provides increased prognostic information above and beyond that provided by pre-existing co-morbidities including age, diabetes mellitus, hypertension and pre-existing cardiovascular disease. Indeed, the incremental risk for death incurred by evidence of myocardial injury appears to be ~5-10x and is amplified by pre-existing cardiovascular disease.

Thus, evidence of myocardial injury has evolved to be a significant (if not the most significant) predictor of mortality among patients admitted to hospital for care of COVID19 disease. It is important to recognize that this elevated morality risk has been identified despite modern and aggressive intensive care therapies including mechanical ventilation, pressor/inotrope therapies and extracorporeal membrane oxygenation (ECMO).

In this context, the investigators propose to evaluate intravenous administration of convalescent plasma (CP) obtained from COVID19 survivors in patients requiring hospitalization for symptomatic "high risk" COVID19 disease as reflected by the presence of elevated hsTPN. Supportive data exist for use of convalescent plasma in the treatment of COVID19 and other overwhelming viral illness. The investigators hypothesize that treatment with COVID19 CP will demonstrate salutary effects on COVID19 disease severity/duration, with the primary objective to reduce mortality and a key secondary objective to reduce the requirement for and/or duration of mechanical ventilation. Finally, as the hospital mortality for patients requiring mechanical ventilation is very high (50 to 80%), these patients will be eligible for COVID19 CP treatment as well, even in the absence of elevated hsTPN. Although considerable overlap of these populations has been observed (elevated hsTPN and requirement for mechanical ventilation) there is not 100% redundancy and it is hopeful that COVID19 CP may provide benefit to these critically ill patients.

This is a single arm, non-randomized, open-label treatment of eligible subjects defined as those who satisfy all inclusion criteria.

Eligible subjects will provide written, informed consent prior to participation. A pregnancy test will be obtained on all women of child-bearing potential. Following informed consent, the following baseline laboratory tests will be obtained:

* Hs-CRP
* D-Dimer
* NT-pro BNP

These laboratory tests which reflect inflammation, thrombosis and myocardial dysfunction (in addition hsTPN which reflects myocardial necrosis) will be repeated every 2 days during hospitalization. Following baseline assessments and informed consent, eligible enrollees will receive convalescent CoVID-19 plasma by intravenous infusion.

COVID-19 Convalescent Plasma Study: Convalescent plasma will be obtained from male donors, nulliparous females, or female donors negative for HLA antibodies at least 28 days following recovery from COVID-19 infection. These donors are used to minimize the risk of transfusion-related acute lung injury (TRALI). Routine ABO and Rh typing and red cell antibody screening will be performed. All plasma will be required to test negative to the following assays per FDA and AABB regulations/ guidelines.

COVID Convalescent Plasma 500 mls will be administered in intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Symptomatic CoVID-19 disease requiring hospitalization
* SARS-CoV-19 PCR positive
* Elevated hsTPN

Exclusion Criteria:

* Multi-organ / system failure
* Renal insufficiency (eGFR <30 or renal replacement therapy)
* Liver dysfunction (>3x ULN SGOT / SGPT)
* Chronic Immunosuppression therapy
* Prior organ transplant
* Prior multiple transfusions for Myelodysplastic syndrome
* Prior treatment with plasma, immunoglobulin transfusion within 30 days
* Allergic reaction to blood/ plasma products
* Pregnant or breast feeding at the time of study
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Reduce mortality | At Day 28
  Reduce mortality of high risk COVID 19 disease compared with historic precedent cohorts (35-50%)

SECONDARY OUTCOMES:
Reduce requirement for mechanical ventilation. | At Day 28
  Reduce the duration of mechanical ventilation in high risk COVID 19 disease compared with historic precedent cohorts (30-60%)
Reduce the duration of mechanical ventilation. | At Day 28
  Reduce the time a participant will remain on the ventilator.
Review of treatment related adverse events. | At Day 28
  Data on the number of participants with treatment related adverse events will be assessed to determine the safety and tolerability of convalescent plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Dean J Kereiakes, MD, Principal Investigator — The Christ Hospital
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No